CLINICAL TRIAL: NCT05250245
Title: Effect of Combined Use of Tolterodine and Continuous Positive Airway Pressure vs Continuous Positive Airway Pressure Only Treatment on Overactive Bladder Symptoms in Women With Moderate-to-severe Obstructive Sleep Apnea Syndrome: A Randomized Clinical Trial
Brief Title: Tolterodine Relieves Overactive Bladder Symptoms in Women With Moderate-to-severe Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Kasım Ertas, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 065
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Overactive Bladder; Obstructive Sleep Apnea; Overactive Bladder Syndrome
MeSH Terms: conditions — Urinary Bladder, Overactive; Sleep Apnea, Obstructive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP only group (Active Comparator): Patients who are going to receive only CPAP treatment for their moderate-to-severe obstructive sleep apnea syndrome (OSAS)
  Interventions: Other: Continuous positive airway pressure therapy (CPAP)
- Combined use of CPAP and tolterodine (Active Comparator): Patients who are going to receive combined use of CPAP and tolterodine 4mg a day treatment for their OSAS
  Interventions: Drug: Tolterodine Tartrate 4 MG; Other: Continuous positive airway pressure therapy (CPAP)

INTERVENTIONS:
Drug: Tolterodine Tartrate 4 MG — Tolterodine is actively being used in the treatment of over active bladder symptoms today
  Arms: Combined use of CPAP and tolterodine
Other: Continuous positive airway pressure therapy (CPAP) — The gold standard for the treatment of confirmed OSAS is continuous positive airway pressure (CPAP) therapy

SUMMARY:
In this study, we aim to determine whether combined tolterodine and CPAP therapy is a more effective treatment for patients with OSAS than CPAP treatment only.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 who underwent polysomnography test with suspicion of OSAS between 01.06.2020-01.01.2022 were enrolled in the study
* Patients with AHI ≥15 (moderate or severe) and OAB-V8≥8 were considered eligible for the study and randomized in two groups to receive either CPAP treatment only or CPAP treatment with tolterodine tartrate

Exclusion Criteria:

* Patients diagnosed with neurological diseases, diabetes mellitus, congestive heart failure, infection, hematuria, urolithiasis, urinary tumors, and urinary retention were excluded from the study. Also, a history of lower urinary tract surgery and medication due to lower urinary tract symptoms were the exclusion criteria.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
OAB-V8 questionnarie score improvement | 3 months
  comparison of the groups in terms of improvements of symptom score questionnaires related to OAB at third month

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yıl University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No